CLINICAL TRIAL: NCT02639104
Title: Could Cervical Postural Changes Affect the Long Thoracic Nerve Electromyographic Findings?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Atilla Kircelli, M.D., Baskent University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KA15-220
Record Dates: First submitted 2015-12-08; First posted 2015-12-24 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Cervicalgia
Keywords: neck pain; cervical lordosis; long thoracic nerve
MeSH Terms: conditions — Neck Pain | interventions — X-Rays; Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cervical postural related neck pain (Experimental): Patients recruit in this group who has a neck pain without radiculopathy. If the patient examination shows neurologic deficits, this patient will exclude in this study. All patients will undergo lateral cervical spine spot radiography and serratus anterior needle electromyography. Cervical segmental angle measurements will be done in all patients.
  Interventions: Radiation: Radiography; Other: Electromyography
- Control group (Sham Comparator): The healthy volunteers recruit in this group. All inviduals will undergo lateral cervical spot radiography and serratus anterior needle electromypography
  Interventions: Radiation: Radiography; Other: Electromyography

INTERVENTIONS:
Radiation: Radiography — Obtaining patients lateral spot cervical spine radiography and will measure;
  1. The segmental angle will be measured from C2-C7 inferior endplates on the lateral radiography
  2. If there is a segmental kyphosis (for example kyphotic angle in C4-5 level), the segmental cobb angle will be measured in the level of the main kyphosis
  3. The segmental cobb angle will be measured between C2-C4 inferior endplates and C4-C7 inferior endplates
Other: Electromyography — Serratus anterior needle electromyography:
  The needle can be inserted into the muscle superficially to the fourth to sixth rib in the medial or posterior axillary line. The usual nerve latency time is between 2.6-4 ms.

SUMMARY:
This study investigates one of the mechanism factors of neck pain. Cervical lordotic angle alterations affect the tension of serratus anterior muscle. Expected result that the long thoracic nerve can be affected in this situation, and could be observed the functional changes of the nerve with serratus anterior electromyographic findings.

DETAILED DESCRIPTION:
Different methods exist in order to evaluate muscle function. For the neck pain, the most commonly used method by researchers and clinicians are spot radiography and surface electromyography (sEMG). Radiographs can be used for the kyphotic angle or cervical lordotic angle measurements. Parameters that can be studied by EMG are amplitude, timing, conduction velocity, fatigability and characteristic frequencies/patterns.

The long thoracic nerve innervates the serratus anterior muscle. This nerve arises from the anterior rami of three spinal nerve roots: the fifth, sixth, and seventh cervical nerves (C5-C7) The nerve descends through the cervicoaxillary canal behind (posterior to) the brachial plexus and the axillary artery and vein, resting on the outer surface of the serratus anterior. The Serratus anterior electromyography, the needle can be inserted into the muscle superficially to the fourth to sixth rib in the medial or posterior axillary line. The usual nerve latency time is between 2.6-4 ms.

In this study, the results of serratus anterior muscle EMG activity and postural cervical angle alterations (lateral radiography) in patients with chronic mechanical neck pain will be compared with healthy volunteers without neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is > to 18 years and <40 yo
* Patient presenting a chronic neck pain (symptoms over 3 months)
* No neurological deficit
* Asymptomatic volunteers (for control group)
* Obtaining the enlightened consent of the patient

Exclusion Criteria:

* Patient having refused to sign his consent
* Patients whose age is < to 18 years or >40 yo.
* Patients with neurologic deficits
* Patients presenting history of allergy
* History of cervical spine surgery
* Patient presenting an anticoagulant or salicylated treatment which can not be interrupted.
* Pregnant woman.
* Patient with acute head and neck trauma
* Patient with a contra-indication to radiography.
* Patient with a psychiatric pathology preventing a clinical evaluation.
* Patient with contra-indication (cutaneous or different) to needle electromyography.
* Surgery contra-indication (cardiac failure, respiratory…)
* Patient without health coverage.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-03 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 1 hour
  Pain is a sensory and emotional experience, modified by multiple factors, including meaning, context, previous pain experience, culture, gender, expectation, anxiety, depression, fear, family and social factors. Patients admitted to hospital experience a high prevalence of moderate and severe pain. The VAS (Visual Analog Scale, 0 mm "no pain", to 100 mm," the worst pain possible ") is used to assess chronic neck pain. The authors aim to find a correlation between factors either neck pain (with VAS), cervical lordosis angle and long thoracic nerve electrophysiological results.

CONTACTS AND LOCATIONS:
Overall Officials: Cem Yılmaz, M.D., Study Director — Baskent University, Department of Neurosurgery
Locations (1):
- Baskent University Konya Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Castelein B, Cools A, Bostyn E, Delemarre J, Lemahieu T, Cagnie B. Analysis of scapular muscle EMG activity in patients with idiopathic neck pain: a systematic review. J Electromyogr Kinesiol. 2015 Apr;25(2):371-86. doi: 10.1016/j.jelekin.2015.01.006. Epub 2015 Jan 31. PMID 25683111